CLINICAL TRIAL: NCT02682797
Title: Use of Spectral Domain Optical Coherence Tomography to Differentiate and Follow-up Senile Retinoschisis and Retinal Detachment
Brief Title: Optical Coherence Tomography Evaluation of Retinoschisis and Retinal Detachment
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Sacu, Assoc. Prof. PD. Dr., Medical University of Vienna
Other Study IDs: 19.08.2015
Record Dates: First submitted 2016-02-05; First posted 2016-02-15 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Retinoschisis
MeSH Terms: conditions — Retinoschisis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: At all study visits a complete ophthalmic examination, visual acuity and refractive error, Spectralis OCT, Cirrus OCT, Topcon OCT, PS-OCT, Optomap Fundus photography will be performed.

SUMMARY:
Retinoschisis is usually a rare self-limited disease and seldom shows progression. There a splitting of the neurosensory retina occurs usually in the inferior temporal. Patients usually have good visual acuity and are asymptomatic. Combination of an inner and outer layer hole is considered high risk factor for development of a schisis detachment. The most important differential diagnosis is an retinal detachment, since if misdiagnosed unnecessary treatment is provided. In clinical examination, both can appear very thin and transparent.

Therefore exact diagnosis of retinoschisis and retinal detachment has to be assessed and regular follow-up controls have to be conducted for sufficient recognition of progression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age.
* Ophthalmoscopic evidence of RS or RD
* Written informed consent has been obtained.

Exclusion Criteria:

* Progression of retinal detachment or retinoschisis requiring surgical treatment
* Contraindication to pupil dilation, known allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 consecutive patients will be recruited for this study; 15 with Retinoschisis and 15 with retinal detachment
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Morphological findings in retinoschisis or retinal detachment in optical coherence tomography scans during follow-up | Baseline
Change or progression of disease measured in optical coherence tomography | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Medical University of Vienna, Austria, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No